CLINICAL TRIAL: NCT03572881
Title: Assessment of Rhythmic Risk in Patients With Type 1 Brugada Syndrome by Pulmonary Infundibulum Mapping
Brief Title: Rhythmic Risk of Type 1 Brugada Syndrome and Pulmonary Infundibulum Mapping
Acronym: SB-CARTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL18_0279
Record Dates: First submitted 2018-06-19; First posted 2018-06-28 (Actual); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Brugada Syndrome Type 1
Keywords: Brugada syndrome; ventricular arrhythmia; sudden death
MeSH Terms: conditions — Brugada Syndrome; Death, Sudden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Asymptomatic (Experimental)
  Interventions: Device: Endocardial mapping
- Symptomatic (Experimental)
  Interventions: Device: Endocardial mapping

INTERVENTIONS:
Device: Endocardial mapping — An endocardial mapping of the pulmonary infundibulum will be performed during the electrophysiological exploration between asymptomatic patients with Brugada type 1 and patients with symptomatic Brugada type 1.

SUMMARY:
Brugada syndrome has been described as the association of a right bundle block with ST segment elevation on the V1 to V3 electrocardiogram in patients with a structurally normal heart. The rhythmic risk is thus difficult to evaluate in asymptomatic patients in whom the rate of events is estimated at 0.2 to 1.4% of events per year. In addition, the predictive value of ventricular pacing remains controversial; There is therefore currently no review to effectively assess rhythmic risk in patients with Brugada type I syndrome.

Investigators aimed to show a difference in pulmonary infundibulum voltage mapping in symptomatic and asymptomatic patients with Brugada type 1 syndrome with a comparable ECG.

The mapping of the pulmonary infundibulum will be performed during electrophysiological exploration. Only the catheter used differs from the usual procedure.

ELIGIBILITY:
Inclusion Criteria:

Group 21

* Brugada Type 1 syndrome
* Age : 50-60 years old
* Asymptomatic
* Signed informed consent

Group2

* Brugada Type 1 syndrome
* Age >18 years old
* Implantable defibrillator
* Having received at least 1 appropriate shock or a sudden sudden death
* Signed informed consent

Groups 1 and 2

Exclusion Criteria:

* Brugada Type 2 or 3 syndrome
* Contraindication to electrophysiological exploration

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Identification of different voltage zones by endocardial mapping of the pulmonary infundibulum between asymptomatic patients with Brugada type 1 and patients with symptomatic Brugada type 1 | Day 1
  The voltage zone are defined with :
  * measurement of unipolar and bipolar local voltage (mV)
  * the scar surface
  * the surface of the bordering area
  * the surface of healthy tissue
  * the quantification of the number of fractionated potentials and density with respect to the size of the infundibulum and the scar (if present)
  * the analysis of the heterogeneity of the voltage (study of dispersion)
  * analysis of propagation card velocities in sinus rhythm and ventricular pacing (mm / s)
  * analysis of ventricular arrhythmia activation if positive ventricular pacing and good hemodynamic tolerance (focal / reentrant / reentrant macro).

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Louis Pradel, Bron, France

IPD SHARING:
Plan to Share IPD: No